CLINICAL TRIAL: NCT05025449
Title: BEFAST (Bubble-Enhanced FAST) for the Evaluation of Solid Organ Injury in Hemodynamically Stable Blunt Abdominal Trauma
Brief Title: BEFAST (Bubble-Enhanced FAST) for the Evaluation of Solid Organ Injury
Acronym: BEFAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laura Oh, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00100619
Record Dates: First submitted 2021-08-26; First posted 2021-08-27 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Abdominal Trauma
Keywords: Ultrasound contrast; Solid organ injury; Blunt abdominal trauma
MeSH Terms: conditions — Abdominal Injuries | interventions — Focused Assessment with Sonography for Trauma

STUDY DESIGN:
Masking Description: The interpretation of the point-of-care emergency medicine (EM) physician (blind to the CT read) will be compared to the interpretations of board-certified radiologists (also blind to the CT read) for the presence or absence of solid organ injury.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Non-enhanced FAST exam followed by BEFAST exam (Experimental): Participants in the emergency department with hemodynamically stable blunt abdominal trauma will receive the standard of care Focused Assessment with Sonography for Trauma (FAST) exam followed by a Bubble-Enhanced FAST exam.
  Interventions: Diagnostic Test: Focused Assessment with Sonography for Trauma (FAST); Drug: Bubble-Enhanced FAST (BEFAST)

INTERVENTIONS:
Diagnostic Test: Focused Assessment with Sonography for Trauma (FAST) — The Focused Assessment with Sonography for Trauma (FAST) exam is widely used and accepted as part of Advanced Trauma Life Support (ATLS) protocol. After consent, a baseline FAST exam will be performed and documented. This FAST will be distinct from the initial ATLS resuscitation FAST in order to avoid any interference in the trauma evaluation. The investigator will use a phased array or curvilinear transducer to record video of their baseline FAST exam.
Drug: Bubble-Enhanced FAST (BEFAST) — Following the FAST exam and using the same machine, a BEFAST exam will be performed using a low mechanical index setting in contrast-specific imaging mode. A 2.4 mL IV dose of Lumason will be injected into the subject's IV, followed by saline flush. The contrast will be injected once for the right side of the body, and once for the left side of the body looking for disruptions in the normal enhancement pattern and evidence of active bleeding. To examine the right side of the body: the liver will be imaged first in arterial phase, followed by the right kidney, before returning to image the liver in venous phase. To examine the left side of the body: the pancreas will be imaged first, followed by the kidney and the spleen. The investigator will note evidence of solid organ injury, free fluid, or active extravasation on both sides of the body; lacerations will be graded by the American Association for the Surgery of Trauma (AAST) criteria.
  Other Names: Lumason

SUMMARY:
The Focused Assessment with Sonography for Trauma (FAST) exam is widely used and accepted as part of advanced trauma life support (ATLS) protocol, but its low sensitivity for identifying solid organ injury in the absence of hemoperitoneum is a significant limitation. Contrast-enhanced ultrasound (CEUS) has the potential to significantly enhance the evaluation of the trauma patient with acute intra-abdominal injury through the use of intravascular microbubbles that allow direct visualization of lacerations to solid organs. European studies have demonstrated that ultrasound contrast markedly improves the sensitivity of ultrasound in detecting solid organ injury, when the exam is performed in the radiology suite. The researchers hypothesize that the bubble-enhanced FAST or BEFAST exam will be more sensitive than traditional FAST for identification of solid organ injury in hemodynamically stable blunt abdominal trauma patients when performed by emergency providers.

DETAILED DESCRIPTION:
Blunt abdominal trauma, whether from motor vehicle crash, assault, fall, or recreational injury, is a leading cause of morbidity and mortality. According to the 2016 National Trauma Database, 12% of all patients with trauma admissions had abdominal trauma, the majority of which is blunt. The diagnosis of intra-abdominal injury due to blunt abdominal trauma can be challenging. The physical exam is unreliable in patients with altered mental status or with impairment due to drugs or alcohol. While computed tomography (CT) can rapidly and accurately diagnose injury, emergency physicians have raised concerns that the use of CT has become overly liberal. The risks of overutilization of CT in hemodynamically stable blunt abdominal trauma include increased health care costs, lengthy stays in the emergency department, risks of contrast-induced nephropathy and radiation-induced malignancy, and patient anxiety when "incidentalomas" are discovered that need extensive and often unnecessary workup.

The Focused Assessment with Sonography for Trauma (FAST) exam is widely used and accepted as part of the advanced trauma life support (ATLS) protocol, but its low sensitivity for identifying solid organ injury in the absence of hemoperitoneum is a significant limitation. Contrast-enhanced ultrasound (CEUS) has the potential to significantly enhance the evaluation of the trauma patient with acute intra-abdominal injury through the use of intravascular microbubbles that allow direct visualization of lacerations to solid organs.

In 2016, the Food and Drug Administration (FDA) approved Lumason (sulfur hexafluoride lipid-type A microsphere) for characterization of focal liver lesions with CEUS in both adult and pediatric patients, opening new areas of research in the United States. Lumason is a second generation contrast agent that is more stable than previous ultrasound contrast agents and does not require refrigeration. Although approved for intravascular and intravesical use, Lumason's use in a trauma exam is off-label in the United States.

After participants provide informed consent, a baseline FAST exam will be performed and documented. This exam will be distinct from the initial ATLS resuscitation FAST in order to avoid any interference in the trauma evaluation. If not already placed, an intravenous line will be established according to standard practice for trauma patients. Following the FAST exam, a bubble-enhanced FAST (BEFAST) exam will be performed using Lumason as the contrast agent. As part of the standard of care, participants will have a CT exam performed within 24 hours, which will provide the gold standard for diagnosis of solid organ trauma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of intra-abdominal injury
* Presentation within 24 hours of injury
* Planned CT of the abdomen/pelvis within 24 hours
* Ability of patient or legally authorized representative to provide informed consent

Exclusion Criteria:

* Co-existing penetrating abdominal injury
* Known hypersensitivity reaction to contrast agent
* Pregnant patients
* Prisoners
* No appropriate IV Line able to be inserted
* Hemodynamic instability at time of enrollment (sustained systolic blood pressure < 90 mm Hg or sustained heart rate (HR) >120 despite initial resuscitation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Oh, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial will be made available for sharing, after de-identification.
Supporting Information: Study Protocol
Time Frame: Data will be made available for sharing beginning 9 months after study publication and ending 36 months after article publication.
Access Criteria: Individual participant data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve the aims in the approved proposal. Proposals should be directed to laura.oh@emory.edu. To gain access, data requestors will need to sign a data use agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Grady Memorial Hospital in Atlanta, Georgia, USA. Participant enrollment began September 30, 2021 and the final study visit occurred on September 14, 2023.
Groups:
- Non-enhanced FAST Exam Followed by BEFAST Exam: Participants in the emergency department with hemodynamically stable blunt abdominal trauma receiving the standard of care Focused Assessment with Sonography for Trauma (FAST) exam followed by a Bubble-Enhanced FAST exam.
  The Focused Assessment with Sonography for Trauma (FAST) exam is widely used and accepted as part of Advanced Trauma Life Support (ATLS) protocol. After consent, a baseline FAST exam is performed and documented. This FAST is distinct from the initial ATLS resuscitation FAST in order to avoid any interference in the trauma evaluation. Following the FAST exam and using the same machine, a BEFAST exam is performed using a low mechanical index setting in contrast-specific imaging mode. A 2.4 mL IV dose of Lumason is injected into the subject's IV, followed by saline flush. The contrast is injected once for the right side of the body, and once for the left side of the body looking for disruptions in the normal enhancement pattern and evidence of active bleeding. To examine the right side of the body: the liver will be imaged first in arterial phase, followed by the right kidney, before returning to image the liver in venous phase. To examine the left side of the body: the pancreas will be imaged first, followed by the kidney and the spleen. The investigator will note evidence of solid organ injury, free fluid, or active extravasation on both sides of the body; lacerations will be graded by AAST criteria.
Period: Overall Study
Arm/Group | Non-enhanced FAST Exam Followed by BEFAST Exam
Started | 267
Completed | 265
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Patient emergently taken to operating room | 1

BASELINE CHARACTERISTICS:
Groups:
- Non-enhanced FAST Exam Followed by BEFAST Exam: Participants in the emergency department with hemodynamically stable blunt abdominal trauma receiving the standard of care Focused Assessment with Sonography for Trauma (FAST) exam followed by a Bubble-Enhanced FAST exam.
Arm/Group | Non-enhanced FAST Exam Followed by BEFAST Exam
Number analyzed (Participants) | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 203
  >=65 years | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 253
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 160
  White | 89
  More than one race | 2
  Unknown or Not Reported | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 267

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Detecting Solid Organ Injury Measured as the Number of True Positives
Description: The performance of the study exams will be assessed as the number of correctly identified solid organ injuries (true positives) detected by FAST exam and BEFAST exam. The presence of injury will be determined by the gold standard of a CT exam, conducted within 24 hours as part of the standard of care.
Time Frame: 1 Day of exam
Population: Two participants were withdrawn from the study after having the FAST exam and before having the BEFAST exam.
Measure: Count of Participants; unit: Participants
Groups:
- Non-enhanced FAST Exam: Participants in the emergency department with hemodynamically stable blunt abdominal trauma receiving the standard of care Focused Assessment with Sonography for Trauma (FAST) exam, followed by a Bubble-Enhanced FAST exam.
- BEFAST Exam: Participants in the emergency department with hemodynamically stable blunt abdominal trauma receiving a Bubble-Enhanced FAST exam, following the standard of care Focused Assessment with Sonography for Trauma (FAST) exam.
Arm/Group | Non-enhanced FAST Exam | BEFAST Exam
Number analyzed (Participants) | 267 | 265
Participants | 18 | 20

2. Primary Outcome: Specificity of Detecting Solid Organ Injury Measured as the Number of True Negatives
Description: The performance of the study exams is assessed as the percentage of correctly identified lack of solid organ injuries (true negatives) detected by FAST and BEFAST exams. The presence of solid organ injury is determined by the gold standard of a CT exam, conducted within 24 hours as part of the standard of care.
Time Frame: 1 Day of exam
Population: Two participants were withdrawn from the study after having the FAST exam and before having the BEFAST exam.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-enhanced FAST Exam | BEFAST Exam
Number analyzed (Participants) | 267 | 265
Participants | 214 | 216

3. Primary Outcome: Number of Enrolled Participants With Successful Exams
Description: The number of successful, completed exams is used to determine whether emergency physicians can incorporate BEFAST evaluation at the point-of-care. The exam is considered complete if the participant tolerates the study without experiencing severe adverse events to contrast and the participant allows the provider to complete the scan, and if the exam results in images of adequate quality to answer the focused clinical question.
Time Frame: 1 Day of exam
Measure: Count of Participants; unit: Participants
Arm/Group | Non-enhanced FAST Exam | BEFAST Exam
Number analyzed (Participants) | 267 | 267
Participants | 263 | 245

4. Primary Outcome: Percent Agreement Between Raters
Description: Emergency physicians' interpretations of the ultrasound exams are compared to interpretations of board-certified radiologists for the presence or absence of solid organ injury, free fluid, or active extravasation. Injured organs are graded per American Association for the Surgery of Trauma (AAST) criteria.
Time Frame: 1 Day of exam
Population: Two participants were withdrawn from the study after having the FAST exam and before having the BEFAST exam.
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Arm/Group | Non-enhanced FAST Exam | BEFAST Exam
Number analyzed (Participants) | 267 | 265
percentage of agreement | 82.6 [77.6 to 86.7] | 76.2 [70.7 to 81.0]

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time of informed consent through completion of both the FAST and BEFAST examinations, on the single day of the study (Day 1). Two participants were withdrawn from the study after having the FAST exam and before having the BEFAST exam.
Arm/Group | Non-enhanced FAST Exam | BEFAST Exam
All-Cause Mortality (participants affected / at risk) | 0/267 | 0/265
Serious Adverse Events (participants affected / at risk) | 0/267 | 0/265
Other Adverse Events (participants affected / at risk) | 0/267 | 2/265
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-enhanced FAST Exam (N=267) | BEFAST Exam (N=265)
Itchy feet (General disorders) | 0 | 1
Nausea (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT05025449/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT05025449/ICF_000.pdf